CLINICAL TRIAL: NCT04448665
Title: The Empiric Antimicrobial Therapy: the Comparison of Initial Clinical Choice of Drugs With the Results of Microbiological Investigations - an Observational Study
Brief Title: Compliance of Initial Empiric Antimicrobial Therapy
Status: Completed | Type: Observational
Sponsor: Military Institute od Medicine National Research Institute (Other)
Responsible Party: Principal Investigator, Dariusz Tomaszewski, MD, PhD, Military Institute od Medicine National Research Institute
Other Study IDs: 681006-08
Record Dates: First submitted 2020-06-23; First posted 2020-06-26 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Anti-Infective Agents
Keywords: empirical therapy; antimicrobial agents; hospital infections
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with suspected infection: The hospitalized patients in whom, based on clinical signs and symptoms, an infection is suspected, and an administration of antimicrobial agents as empiric therapy is necessary.
  Interventions: Diagnostic Test: microbiological investigation

INTERVENTIONS:
Diagnostic Test: microbiological investigation — a microbiological tests, including isolation of the pathogen and analysis of their susceptibility/resistance to antimicrobial agents

SUMMARY:
Hospital infections comprise about half of all undesirable complications related to hospital treatment. In case of bacterial infection administration of antimicrobial agent is a therapy of choice. For maximum effectiveness, antimicrobial agents should be administered quickly in optimal doses. Moreover, the therapeutic concentration of properly selected drugs should be achieved as soon as possible. The relation between delays in the administration of antibiotics and increased mortality is well known. That is why proper empiric therapy is so important. Before antimicrobial investigation is completed, which may last up to 72 hours, a wide-spectrum antimicrobial should be administered according to the type of infection, its origin, and the characteristics of the local pathogens.

The objective of this study is to compare the initial choice of empiric antimicrobial therapy and the results of both microbiological identification and susceptibility/resistance analysis of isolated pathogens.

This project was designed as a prospective cohort study. Analysis was performed in a large multidisciplinary academic hospital and trauma center. All decisions on empiric therapy with antimicrobial used in infections caused by multidrug-resistant pathogens, that are made in different hospital wards except intensive care, are required by hospital procedures to be confirmed by intensivists. In our analysis, the initial choice of empiric therapy in the hospital wards other than the critical care unit was compared with the results of microbiological investigations and susceptibility/resistance analyses of isolated pathogens.

Accurate microbial identification was performed with a VITEK® 2 automatic testing system. The microbroth dilution method with VITEK® 2 AST cards was used for the antibiotic susceptibility testing of isolated pathogens.

Microbiological analyses were performed between 2018 and 2020 according to the regulations of the European Committee on Antimicrobial Susceptibility (EUCAST, version 9.0, 2019) and the National Reference Centre for Susceptibility Testing (NRCST, Warsaw, Poland).

ELIGIBILITY:
Eligibility Criteria:

- all patients in whom, based on clinical signs and symptoms, an infection is suspected, and an administration of antimicrobial agents as empiric therapy was necessary

Eclusion Criteria:

- none.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Due to study design we performed no descriptive analyses of the study population.
Sampling Method: Non-Probability Sample
Enrollment: 267 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
Accuracy of initial empiric therapy | Immediately after the completion of microbiological analyses
  The comparison of initially administered antimicrobial agent with the results of microbiological analyses (susceptibility/resistance of the isolated pathogen).

CONTACTS AND LOCATIONS:
Overall Officials: Dariusz Tomaszewski, MD, PhD, Study Director — Department of Anesthesiology and Intensive Therapy
Locations (1):
- Department of Anesthesiology and Intensive Therapy, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided